CLINICAL TRIAL: NCT04772196
Title: Temporal Profile of Serum Vitamin D Levels and Outcomes After Total Ankle Arthroplasty, Ankle Arthrodesis and First Metatarsophalangeal Joint Arthrodesis
Brief Title: Temporal Profile of Serum Vitamin D Levels in Foot and Ankle Fusion Surgery
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Prisma Health-Midlands (Other)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00095065
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Ankle Arthrodesis; MTP Arthrodesis
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either standard of care or supplemental Vitamin D3 following total ankle arthroplasty, ankle arthrodesis, or first metatarsophalangeal joint arthrodesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Group (No Intervention): Patients enrolled in the control group will receive standard of care.
- Vitamin D Supplementation Group (Experimental): Patients enrolled in the Vitamin D Supplementation Group will receive 50,000 IU Vitamin D3 weekly for 8 weeks.
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — 50,000 IU Vitamin D3 weekly for 8 weeks
  Arms: Vitamin D Supplementation Group

SUMMARY:
Vitamin D is important for bone health and recent research has emphasized the importance of adequate vitamin D levels for bone healing, wound healing, and possibly preventing infections post-operatively. This study will assess the effect of vitamin D supplementation on patient outcomes following ankle arthrodesis or first metatarsophalangeal joint arthrodesis.

DETAILED DESCRIPTION:
The current status of knowledge includes preliminary research correlating hypovitaminosis, or low vitamin D status, to worse outcomes. In orthopaedic patients, vitamin D deficiency is prevalent among those scheduled to undergo surgery.

Vitamin D is important for calcium homeostasis and bone health, as well as for activation and differentiation of macrophages, dendritic cells, and lymphocytes. A recent retrospective review of outcomes in revision total joint arthroplasty patients showed that patients with low vitamin D had higher rates of postoperative complications and periprosthetic infections. Additionally, another retrospective study correlated low vitamin D levels with lower patient reported outcomes (PROs) after total hip arthroplasty. Current retrospective studies suggest that having low vitamin D levels may lead to impaired fracture healing, increased wound complication rates, and a higher risk of infections.

Given this background information, this study will investigate a series of patients undergoing ankle arthrodesis and first metatarsophalangeal joint (MTP) arthrodesis. Our study will serve to enhance the current knowledge as a level 1 randomized control study on the effect of Vitamin D supplementation on the complication rate following these two arthrodesis procedures. Our endpoints for complications will be defined as infection, wound healing complications, need for readmission, need for re-operation and nonunion as evidenced clinically and radiographically.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age
* Subject is undergoing ankle arthrodesis or MTP arthrodesis
* Subject speaks and understands English

Exclusion Criteria:

* Subject is < 18 years of age
* Subject has an active joint infection
* Subject is unable to provide consent
* Subject is a prisoner

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Post-surgical complication rate following Vitamin D3 supplementation | 6 months
  Patients will be followed for 6 months post-operatively to determine overall complication rate in patients receiving Vitamin D3 supplementation vs. standard of care. Complications will include infection, wound healing complications, readmission, re-operation, and clinical or radiographic nonunion.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bentli R, Taskapan H, Toktas H, Ulutas O, Ozkahraman A, Comert M. Significant independent predictors of vitamin d deficiency in inpatients and outpatients of a nephrology unit. Int J Endocrinol. 2013;2013:237869. doi: 10.1155/2013/237869. Epub 2013 May 12. PMID 23737771
- [Background] Bogunovic L, Kim AD, Beamer BS, Nguyen J, Lane JM. Hypovitaminosis D in patients scheduled to undergo orthopaedic surgery: a single-center analysis. J Bone Joint Surg Am. 2010 Oct 6;92(13):2300-4. doi: 10.2106/JBJS.I.01231. PMID 20926724
- [Background] Hewison M. Vitamin D and the immune system: new perspectives on an old theme. Endocrinol Metab Clin North Am. 2010 Jun;39(2):365-79, table of contents. doi: 10.1016/j.ecl.2010.02.010. PMID 20511058
- [Background] Lavernia CJ, Villa JM, Iacobelli DA, Rossi MD. Vitamin D insufficiency in patients with THA: prevalence and effects on outcome. Clin Orthop Relat Res. 2014 Feb;472(2):681-6. doi: 10.1007/s11999-013-3172-7. PMID 23868422
- [Background] Somerson JS, Bartush KC, Shroff JB, Bhandari M, Zelle BA. Loss to follow-up in orthopaedic clinical trials: a systematic review. Int Orthop. 2016 Nov;40(11):2213-2219. doi: 10.1007/s00264-016-3212-5. Epub 2016 May 3. PMID 27142421
- [Background] Zelle BA, Bhandari M, Sanchez AI, Probst C, Pape HC. Loss of follow-up in orthopaedic trauma: is 80% follow-up still acceptable? J Orthop Trauma. 2013 Mar;27(3):177-81. doi: 10.1097/BOT.0b013e31825cf367. PMID 23449099
- [Background] Kristman V, Manno M, Cote P. Loss to follow-up in cohort studies: how much is too much? Eur J Epidemiol. 2004;19(8):751-60. doi: 10.1023/b:ejep.0000036568.02655.f8. PMID 15469032
- [Background] Nwankwo EC Jr, Labaran LA, Athas V, Olson S, Adams SB. Pathogenesis of Posttraumatic Osteoarthritis of the Ankle. Orthop Clin North Am. 2019 Oct;50(4):529-537. doi: 10.1016/j.ocl.2019.05.008. PMID 31466668